CLINICAL TRIAL: NCT00890474
Title: Moxibustion for Fetus in Breech Presentation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss National Science Foundation (Other); Loterie Romande (Unknown)
Responsible Party: Marie-Julia Guittier, Hôpitaux Universitaires de Genève
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Moxibustion_siege
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Breech Presentation
Keywords: Breech presentation at 34 to 36 weeks of gestation
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxibustion (Experimental)
  Interventions: Procedure: Moxibustion of the BL67 acupoint
- Control (No Intervention)

INTERVENTIONS:
Procedure: Moxibustion of the BL67 acupoint — Moxibustion sessions every day (every other day in hospital, self-administration at home the other day) during a maximum of 14 days. Stopped if cephalic version.
  Arms: Moxibustion

SUMMARY:
Objective: To evaluate moxibustion of the BL67 acupoint between 34 and 38 weeks of gestation to facilitate cephalic version of breech presentation in a Western setting. The hypothesis is that moxibustion increase the likelihood of cephalic version.

Design: Randomised controlled trial Setting: University hospital. Population: A total of 212 consenting women between 34 and 36 weeks of gestation with a single fetus in breech presentation will be randomised to moxibustion (n=106) or expectant management (n=106).

Main Outcome Measure: Cephalic presentation at delivery or before external cephalic version.

ELIGIBILITY:
Inclusion Criteria:

* Breech presentation
* 34 to 36 weeks of gestation
* Single fetus

Exclusion Criteria:

* Uterine malformation
* Placenta praevia
* Transverse lie

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2004-10; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Cephalic presentation at delivery or before external cephalic version | end of pregnancy

SECONDARY OUTCOMES:
Mode of delivery | end of pregnancy
Women's views on the intervention | end of pregnancy
External cephalic version | end of pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

REFERENCES:
- [Derived] Guittier MJ, Pichon M, Dong H, Irion O, Boulvain M. Moxibustion for breech version: a randomized controlled trial. Obstet Gynecol. 2009 Nov;114(5):1034-1040. doi: 10.1097/AOG.0b013e3181bc707a. PMID 20168104